CLINICAL TRIAL: NCT00132639
Title: Randomized Phase II Study of the Induction Chemotherapy With Docetaxel Alone vs CDDP + Docetaxel for C-stage IB-II Non-Small Cell Lung Cancer (JCOG 0204-MF)
Brief Title: Study of Preoperative Docetaxel or Cisplatin (CDDP) + Docetaxel for C-stage IB-II Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG 0204-MF; C000000032
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Neoplasms
Keywords: pulmonary neoplasm; preoperative chemotherapy; cisplatin, docetaxel; randomized trial; clinical stage IB or II nonsmall cell lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Preoperative docetaxel-cisplatin combination chemotherapy
  Interventions: Drug: Preoperative docetaxel-cisplatin combination chemotherapy
- 2 (Active Comparator): Preoperative docetaxel monotherapy
  Interventions: Drug: Preoperative docetaxel monotherapy

INTERVENTIONS:
Drug: Preoperative docetaxel-cisplatin combination chemotherapy — Preoperative docetaxel-cisplatin combination chemotherapy
  Arms: 1
Drug: Preoperative docetaxel monotherapy — Preoperative docetaxel monotherapy
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the preoperative docetaxel and docetaxel-cisplatin combination in c-stage IB/II NSCLC, and select the optimal preoperative therapy for phase III trials.

DETAILED DESCRIPTION:
Preoperative chemotherapy has substantial theoretical advantage. Several controlled trials are under way in early stage (clinical stage IB-II) nonsmall cell lung cancer (NSCLC). In each trial, platinum-based doublet chemotherapy is employed. Although platinum-based doublet is the treatment of choice for advanced NSCLC, risk/benefit balance might well be different in earlier stages. There have been no prospective randomized trials to choose an optimal preoperative chemotherapy in early stage NSCLC.

Comparison: Preoperative cisplatin-docetaxel combination versus docetaxel monotherapy in clinical stage IB/II NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, pathologically documented NSCLC
* Clinical stages IB (T2N0M0), IIA (T1N1M0) or IIB (T2N1M0 or T3N0M0)
* Ages: 15-74 years old
* ECOG performance status 0 or 1
* Measurable disease
* Ample organ function
* Signed informed consent

Exclusion Criteria:

* Invasion to the first rib or more superior chest wall
* Metastasis to, or involvement of, mediastinal node
* Active concomitant malignancy
* Unstable angina, recent myocardial infarction, or heart failure
* Uncontrolled diabetes or hypertension
* Pregnant or lactating women
* Other severe complications
* Systemic use of corticosteroids

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
disease-free survival rate at 1 year | during the study conduct

SECONDARY OUTCOMES:
overall survival | during the study conduct
disease-free survival | during the study conduct
treatment compliance | during the study conduct
response rate to chemotherapy | during the study conduct
pathologic complete response (CR) rate | during the study conduct
complete resection rate | during the study conduct
post-surgical morbidity/mortality | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Harubumi Kato, MD, PhD, Study Chair — Tokyo Medical University
Locations (1):
- National Cancer Center, Chuo-ku,Tsukiji,5-1-1, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.jcog.jp/